CLINICAL TRIAL: NCT00960193
Title: A One-Directional, Open-Label Drug-Food Interaction Study to Investigate the Effects of Multiple-Daily Consumptions of Seville Orange Juice on the Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Food Interaction Study of Seville Orange Juice and Colchicine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1018
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: blood levels over time; colchicine; seville orange juice; pharmacokinetics
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine Alone (Active Comparator): baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Seville Orange Juice (Experimental): colchicine pharmacokinetics in presence of Seville orange juice
  Interventions: Drug: Colchicine; Other: Seville Orange Juice

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone in the morning on Day 1 and a single dose of 0.6 mg colchicine administered with Seville orange juice in the morning on Day 18 after an overnight fast of at least 10 hours.
Other: Seville Orange Juice — 240 mL of Seville orange juice administered in the morning and evening on Days 15 to 18.
  Arms: Colchicine with Seville Orange Juice

SUMMARY:
Seville orange juice is an inhibitor of the intestinal cytochrome P450 (CYP) 3A4 enzyme, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple daily consumptions of Seville orange juice on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Seville orange juice is an inhibitor of the intestinal cytochrome P450 (CYP) 3A4 enzyme, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple daily consumptions of Seville orange juice on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. Twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one dose of colchicine (1 x 0.6 mg tablet) on Day 1, after an overnight fast. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose to adequately define the baseline pharmacokinetics of colchicine. After a 14 day washout period, starting on the morning of Day 15 and continuing through Day 17, subjects will return to the clinic for consumption of an administered 240 ml dose of Seville orange juice in the morning and evening. At 8am on Day 18 after an overnight fast, all subjects will receive a co-administered single oral dose of colchicine (1 x 0.6 mg) and Seville orange juice (1 x 240 ml). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose to adequately define the pharmacokinetics of colchicine in the presence of Seville orange juice. Subjects will consume the final administered 240 ml dose of Seville orange juice in the evening on Day 18. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to dosing and at approximately 1, 2, and 3 hours following drug administration on Days 1 and 18 to coincide with peak plasma concentrations of colchicine. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive
* Hemoglobin greater than or equal to 11.5g/dL

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine
* Intolerance or food allergy to Seville orange juice

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Wason S, DiGiacinto JL, Davis MW. Effects of grapefruit and Seville orange juices on the pharmacokinetic properties of colchicine in healthy subjects. Clin Ther. 2012 Oct;34(10):2161-73. doi: 10.1016/j.clinthera.2012.08.007. Epub 2012 Aug 31. PMID 22940371
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Colchicine Alone, Colchicine With Seville Orange Juice: On the morning of Day 1, subjects received a single dose of colchicine 0.6 mg after an overnight fast, followed by a 14 day washout period. On Days 15-17, each subject received one 240 ml serving of Seville orange juice in the morning and evening. On Day 18, subjects received one dose of colchicine 0.6 mg in the morning along with a 240 ml serving of Seville orange juice. Subjects received a final 240 ml serving of Seville orange juice in the evening on Day 18.
Period: Colchicine Alone
Arm/Group | Colchicine Alone, Colchicine With Seville Orange Juice
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone, Colchicine With Seville Orange Juice
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Seville Orange Juice Alone
Arm/Group | Colchicine Alone, Colchicine With Seville Orange Juice
Started | 23
Completed | 23
Not Completed | 0
Period: Colchicine With Seville Orange Juice
Arm/Group | Colchicine Alone, Colchicine With Seville Orange Juice
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone, Colchicine With Seville Orange Juice
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.83 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Colchicine
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to colchicine dosing on Days 1 and 18, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hours after colchicine dose administration.
Population: 24 subjects were enrolled in this study. One subject was withdrawn due to failure to arrive for the Day 15 orange juice dose.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 after an overnight fast, followed by a washout period of 14 days.
- Colchicine With Seville Orange Juice: On Days 15 to 17, each subject received one 240 ml serving of Seville orange juice in the morning and evening. Then, on Day 18, each subject received one 0.6 mg colchicine tablet and one 240 ml serving of Seville orange juice in the morning after an overnight fast. A final 240 ml serving of Seville orange juice was administered in the evening on Day 18.
Arm/Group | Colchicine Alone | Colchicine With Seville Orange Juice
Number analyzed (Participants) | 23 | 23
pg/mL | 2,328.44 (980.15) | 1,668.33 (423.36)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Colchicine Alone | Colchicine With Seville Orange Juice
Number analyzed (Participants) | 23 | 23
pg*hr/mL | 10,261.93 (4,307.62) | 7,634.86 (2,678.60)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: 24 subjects were enrolled in this study. One subject was withdrawn due to failure to arrive for the Day 15 orange juice dose. The pharmacokinetic parameter, AUC(0-∞), could not be determined for 1 subject in the Colchicine Alone group and for 2 subjects in the Colchicine with Seville orange juice group.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Colchicine Alone | Colchicine With Seville Orange Juice
Number analyzed (Participants) | 22 | 21
pg*hr/mL | 12,071.30 (4,657.94) | 9,148.05 (2,743.54)

ADVERSE EVENTS:
Description: 24 subjects were enrolled in this study. One subject was withdrawn from the study due to failure to arrive for the Day 15 Seville orange juice dose.
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at after an overnight fast, followed by a washout period of 14 days.
- Seville Orange Juice Alone: On Days 15 to 17, each subject received one 240 ml serving of Seville orange juice in the morning and evening.
- Colchicine With Seville Orange Juice: On Day 18, each subject received one 0.6 mg colchicine tablet and one 240 ml serving of Seville orange juice after an overnight fast. A final 240 ml serving of Seville orange juice was administered in the evening on Day 18.
Arm/Group | Colchicine Alone | Seville Orange Juice Alone | Colchicine With Seville Orange Juice
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 5/24 | 0/23 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Alone (N=24) | Seville Orange Juice Alone (N=23) | Colchicine With Seville Orange Juice (N=23)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days